CLINICAL TRIAL: NCT03486223
Title: Effect of Inhibition Soluble Epoxide Hydrolase on Insulin Sensitivity in Humans
Brief Title: Soluble Epoxide Hydrolase Inhibition and Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Matt Luther, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 170468; 5R01DK117875 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; PreDiabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Prediabetic State; Obesity | interventions — N-((4-cyano-2-(trifluoromethyl)phenyl)methyl)-3-((4-methyl-6-(methylamino)-1,3,5-triazin-2-yl)amino)cyclohexanecarboxamide

STUDY DESIGN:
Intervention Model Description: Arm 1 and 2 are crossover arms
Who Masked: Participant, Investigator
Masking Description: Arms 1/2 are placebo controlled and blinded to investigator and participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then GSK2256294 (Experimental): Subjects will receive placebo oral capsule daily by mouth for 7 days, then seven week washout and then GSK2256294 daily by mouth for 7 days.
  Interventions: Drug: GSK2256294; Drug: Placebo oral capsule
- GSK2256294 then Placebo (Experimental): Subjects will receive GSK2256294 daily by mouth for 7 days, then seven week washout and then placebo oral capsule daily by mouth for 7 days.
  Interventions: Drug: GSK2256294; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: GSK2256294 — Drug will be taken daily by mouth for 7 days.
  Other Names: GSK2256294 10mg oral capsule
Drug: Placebo oral capsule — Placebo will be taken daily by mouth for 7 days.
  Other Names: Placebo

SUMMARY:
The purpose of this study is to test how soluble epoxide hydrolase (sEH) inhibition with GSK2256294 affects tissue sEH activity and insulin sensitivity.

DETAILED DESCRIPTION:
We will test the hypothesis that soluble epoxide hydrolase (sEH) inhibition with GSK2256294 improves insulin sensitivity using the gold-standard, hyperinsulinemic-euglycemic clamps, with stable isotope dilution to assess hepatic gluconeogenesis. We will assess insulin-stimulated vasodilation in the forearm using plethysmography and in the renal vasculature using para-aminohippurate (PAH, IND#133828) clearance. We will obtain adipose and muscle tissue before and after clamp to assess insulin signaling in these tissues.

Subjects are randomized to treatment with the sEH inhibitor GSK2256294 (10mg/day) or matching placebo for one week. On the seventh day of drug treatment, subjects will report to the CRC in the morning after an overnight fast to undergo a hyperinsulinemic-euglycemic clamp with adipose tissue biopsies.

During the Hyperinsulinemic-euglycemic clamp, insulin will be infused for 2 hours at low dose (20 mU/m2/min) and 2 hours at high dose (80 mU/m2/min) to assess insulin sensitivity. The Glucose Infusion Rate (GIR) will be adjusted to maintain glucose near 95 mg/dL. The average GIR during the final 30 minutes of the high dose period will be used as the measure of insulin sensitivity.

After completion of the study day, subjects will undergo a seven-week washout from study drug and then receive the opposite drug for one week. On the seventh day of treatment they will report to the CRC after an overnight fast and repeat the study day protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women,
2. Age 21 to 50 years, and
3. Pre-diabetes as defined by

   1. Fasting plasma glucose 100-125 mg/dL, or
   2. Two-hour plasma glucose 140-199 mg/dL, or
   3. HbA1c 5.7-6.4%
4. BMI ≥ 30 kg/m2, inclusive
5. For female subjects, the following conditions must be met:

   1. Postmenopausal status for at least one year, or
   2. Status-post surgical sterilization, or
   3. If of childbearing potential, utilization of adequate birth control and willingness to undergo serum β-hcg testing prior to drug treatment and on every study day.

Exclusion Criteria:

1. Diabetes type 1 or type 2, as defined by a fasting plasma glucose of 126 mg/dL or greater, a two-hour plasma glucose of 200 mg/dL or greater, a HbA1c >6.4%, or the use of anti-diabetic medication
2. Subjects who have participated in a weight-reduction program during the last six month or whose weight has increased or decreased more than two kg over the preceding six months
3. Resistant hypertension, defined as hypertension requiring the administration of more than three anti-hypertensive agents including a diuretic to achieve control
4. Use of spironolactone
5. Pregnancy or breast-feeding
6. Any history of smoking
7. Any history of cancer including skin cancer, any history of a precancerous lesion, abnormal PSA, or lack of screening adherent to American Cancer Society Guidelines for the Early Detection of Cancer
8. Cardiovascular disease such as myocardial infarction within six months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep-vein thrombosis, pulmonary embolism, second- or third-degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
9. Abnormal corrected QT interval on screening ECG (QTc).
10. Treatment with anticoagulants
11. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
12. History or presence of immunological or hematological disorders
13. Diagnosis of asthma requiring regular inhaler use
14. Clinically significant gastrointestinal impairment that could interfere with drug absorption
15. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >3.0 x upper limit of normal range)
16. History of gastrointestinal bleed
17. Estimated glomerular filtration rate (eGFR)<60 mL/min/1.73 m2 or with an albumin-to-creatinine ratio (UACR) >300µg/mg, where eGFR is determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine is expressed in mg/dL and age in years: eGFR (mL/min/1.73m2)=186 • Scr-1.154 • age-0.203 • (1.212 if black) • (0.742 if female)
18. Hematocrit <35%
19. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
20. Treatment with chronic systemic glucocorticoid therapy
21. Treatment with lithium salts
22. History of alcohol or drug abuse
23. Treatment with any investigational drug in the month preceding the study
24. Mental conditions rendering a subject unable to understand the nature, scope, and possible consequences of the study
25. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Luther, MD, Principal Investigator — Vanderbilt University Medical Center; Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Available upon request.

REFERENCES:
- [Background] Luther JM, Brown NJ. Epoxyeicosatrienoic acids and glucose homeostasis in mice and men. Prostaglandins Other Lipid Mediat. 2016 Sep;125:2-7. doi: 10.1016/j.prostaglandins.2016.07.010. Epub 2016 Jul 19. PMID 27448715
- [Background] Gangadhariah MH, Dieckmann BW, Lantier L, Kang L, Wasserman DH, Chiusa M, Caskey CF, Dickerson J, Luo P, Gamboa JL, Capdevila JH, Imig JD, Yu C, Pozzi A, Luther JM. Cytochrome P450 epoxygenase-derived epoxyeicosatrienoic acids contribute to insulin sensitivity in mice and in humans. Diabetologia. 2017 Jun;60(6):1066-1075. doi: 10.1007/s00125-017-4260-0. Epub 2017 Mar 28. PMID 28352940
- [Background] Ramirez CE, Shuey MM, Milne GL, Gilbert K, Hui N, Yu C, Luther JM, Brown NJ. Arg287Gln variant of EPHX2 and epoxyeicosatrienoic acids are associated with insulin sensitivity in humans. Prostaglandins Other Lipid Mediat. 2014 Oct;113-115:38-44. doi: 10.1016/j.prostaglandins.2014.08.001. Epub 2014 Aug 28. PMID 25173047
- [Result] Luther JM, Ray J, Wei D, Koethe JR, Hannah L, DeMatteo A, Manning R, Terker AS, Peng D, Nian H, Yu C, Mashayekhi M, Gamboa J, Brown NJ. GSK2256294 Decreases sEH (Soluble Epoxide Hydrolase) Activity in Plasma, Muscle, and Adipose and Reduces F2-Isoprostanes but Does Not Alter Insulin Sensitivity in Humans. Hypertension. 2021 Sep;78(4):1092-1102. doi: 10.1161/HYPERTENSIONAHA.121.17659. Epub 2021 Aug 30. PMID 34455816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 volunteers were screened for inclusion
Pre-assignment Details: 16 individuals were randomized. Of those not randomized, 19 did not meet inclusion criteria and were excluded. 1 participant was randomized but was excluded due to illness prior to receiving any study intervention.
Period: Intervention 1
Arm/Group | Placebo Then GSK2256294 | GSK2256294 Then Placebo
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — received oral steroids for sinus infection; randomized but did not receive intervention | 0 | 1
Period: Washout
Arm/Group | Placebo Then GSK2256294 | GSK2256294 Then Placebo
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Placebo Then GSK2256294 | GSK2256294 Then Placebo
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant included here (in GSK-then-placebo arm) was randomized but did not receive intervention or complete a study day
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then GSK2256294 | GSK2256294 Then Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (8) | 48 (10) | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 6 | 11
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Glucose [Mean (Standard Deviation); unit: mg/dl] | 97 (8) | 96 (8) | 97 (8)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 39 (7) | 43 (9) | 41 (8)
Waist circumference [Mean (Standard Deviation); unit: cm] | 112 (14) | 121 (24) | 116 (20)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 50 (11) | 47 (7) | 48 (9)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 117 (48) | 128 (65) | 122 (55)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity determined by Hyperinsulinemic-Euglycemic Clamp as the glucose infusion rate (GIR) per fat-free-mass (FFM) during high dose insulin infusion
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: mg/kg/FFM/min
Groups:
- Placebo: Placebo oral capsule: Placebo will be taken daily by mouth for 7 days.
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
mg/kg/FFM/min | 12.0 (4.3) | 11.6 (3.7)
Statistical Analysis 1: Comparison: Placebo vs GSK2256294; A sample size of 16 per group was estimated to have 86% power to detect a within-subject difference of 3.76 (80% of the above difference) or larger (with an SD for the within-subject difference of 4.6) in insulin sensitivity; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney) — Wilcoxon signed-rank test was used for the within-subject comparison of GSK2256294 versus placebo

2. Secondary Outcome: Forearm Blood Flow (FBF)
Description: Insulin stimulated forearm blood flow determined by strain-gauge plethysmography
Time Frame: Day 7
Population: Unable to obtain FBF measurement during 2 Placebo study days
Measure: Mean (Standard Deviation); unit: ml/min/100ml
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 13 | 15
ml/min/100ml | 3.5 (1.9) | 3.1 (1.2)

3. Secondary Outcome: Insulin Signaling in Tissue
Description: Insulin stimulated phosphorylated AKT to total AKT ratio (pAKT/AKT) in adipose and muscle tissue sample. AKT is an insulin sensitive serine/threonine kinase also known as protein kinase B.
Time Frame: Day 7
Population: Unable to obtain adipose sample for pAKT measurement during 2 Placebo study days
Measure: Mean (Standard Deviation); unit: pAKT/pAKT ratio
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 13 | 15
pAKT/pAKT ratio
  Adipose Tissue | 0.21 (0.14) | 0.19 (0.18)
  Muscle Tissue | 0.74 (0.55) | 0.73 (0.58)

4. Secondary Outcome: Blood Pressure
Description: determined by non-invasive brachial blood pressure measurement (systolic blood pressure, SBP; diastolic blood pressure, DBP)
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
mmHg
  SBP | 122.9 (11.0) | 124.3 (9.6)
  DBP | 77.4 (6.8) | 78.9 (8.7)

5. Other Pre Specified Outcome: Soluble Epoxide Hydrolase Activity
Description: soluble epoxide hydrolase (sEH) activity measured by 14,15-DHET conversion rate in plasma
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pmol 14,15-DHET/ml/hr
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
pmol 14,15-DHET/ml/hr | 4.1 (4.5) | 1.9 (2.6)

6. Secondary Outcome: Renal Plasma Flow (RPF)
Description: Renal plasma flow determined by PAH infusion, ml/min/per 1.73 m^2 body surface area
Time Frame: Day 7
Population: Unable to obtain RBF measurement in 8 participants due to availability of PAH
Measure: Mean (Standard Deviation); unit: ml/min/per 1.73 m^2
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 7 | 8
ml/min/per 1.73 m^2 | 648 (138) | 614 (103)

7. Other Pre Specified Outcome: Plasma Total Epoxyeicosatrienoic Acids (EETs)
Description: total Epoxyeicosatrienoic acids in plasma
Time Frame: Day 7
Population: Adequate sample not available in 1 participant during GSK
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 14
pmol/mL | 21.4 (8.4) | 22.4 (9.3)

8. Other Pre Specified Outcome: Plasma IL-6
Description: Plasma cytokine interleukin-6 (IL-6)
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pmol/ml
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
pmol/ml | 1.48 (0.61) | 1.48 (0.69)

9. Other Pre Specified Outcome: Plasma VEGF
Description: Plasma vascular endothelial growth factor (VEGF)
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
pg/ml | 31.9 (18.6) | 29.0 (24.4)

10. Other Pre Specified Outcome: Adipose Tissue Total Epoxyeicosatrienoic Acids (EETs)
Description: total Epoxyeicosatrienoic acids in adipose tissue (pmol per mg tissue)
Time Frame: Day 7
Population: Adequate sample not available in 1 participant during GSK
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 14
pmol/mg | 176 (291) | 66 (44)

11. Other Pre Specified Outcome: Soluble Epoxide Hydrolase Activity in Tissue
Description: soluble epoxide hydrolase (sEH) activity measured by 14,15-DHET conversion rate in adipose and muscle, per mg tissue
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pmol 14,15-DHET/mg tissue/hr
Arm/Group | Placebo | GSK2256294
Number analyzed (Participants) | 15 | 15
pmol 14,15-DHET/mg tissue/hr
  Adipose | 2176 (965) | 1280 (675)
  Muscle | 3.5 (1.6) | 1.9 (1.1)

ADVERSE EVENTS:
Time Frame: Baseline to one month post-intervention (approximately 3 months)
Arm/Group | Placebo | GSK2256294
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | GSK2256294 (N=15)
Flushing (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Increased frequency of bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia of lips (Nervous system disorders) | 1 (1) | 0 (0)
Rash at biopsy dressing site (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Increased thirst (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was not sufficient for subgroup analysis for race and gender, due to drug expiration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03486223/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03486223/SAP_003.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03486223/ICF_004.pdf